CLINICAL TRIAL: NCT03601169
Title: Comparison of MMFS Dosages for Improving Cognition, Mood, and Sleep Quality in Older Adults
Brief Title: Comparison of MMFS Dosages in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NC010
Record Dates: First submitted 2018-07-05; First posted 2018-07-26 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Anxiety; Depression; Sleep Quality; Cognitive Impairment
Keywords: cognition; mood; sleep
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction | interventions — threonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose MMFS-205-SR (Experimental): Low dose, oral MMFS-205-SR twice daily (1,000 or 1,500 mg/day total, depending on lean body mass: ~22mg/kg LBM/day) for 6 weeks
  Interventions: Dietary Supplement: Low Dose MMFS-205-SR
- High Dose MMFS-205-SR (Experimental): High dose, oral MMFS-205-SR twice daily (1,500 or 2,000 mg/day total, depending on lean body mass: ~33mg/kg LBM/day) for 6 weeks
  Interventions: Dietary Supplement: High Dose MMFS-205-SR
- Placebo (Placebo Comparator): Oral inactive placebo twice daily for 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low Dose MMFS-205-SR — Twice daily, oral 500mg tablets
  Other Names: L-threonic acid magnesium salt, L-TAMS
  Arms: Low Dose MMFS-205-SR
Dietary Supplement: High Dose MMFS-205-SR — Twice daily, oral 500mg tablets
  Other Names: L-threonic acid magnesium salt, L-TAMS
  Arms: High Dose MMFS-205-SR
Dietary Supplement: Placebo — Twice daily, oral
  Other Names: inactive sugar pill
  Arms: Placebo

SUMMARY:
This study is designed to compare the effectiveness of different doses of brain health supplement MMFS relative to placebo on cognition, mood, and sleep quality.

DETAILED DESCRIPTION:
This is a phase 2 study in older adults with at least mild progressive behavioral symptoms, subjective sleep maintenance problems, and at least mild progressive cognitive deficit. The study is a randomized, double-blind, placebo-controlled, three-way crossover design, in which participants will receive oral placebo, low dose MMFS, and high dose MMFS twice daily for 6 weeks. Over three study periods (2 weeks each), subjects will receive two different dosages of MMFS (low dose: ~22.5 mg/kg LBM/day and high dose: ~35 mg/kg LBM/day) and placebo. After periods 1 and 2 there will be a one week washout period in which the subject will not take any study tablets. Randomized patients and their informants (required) will complete 5 assessments total: at baseline in the clinic (visit 1; prior to taking any study tablets), and 4 times at home via online assessments (at the beginning of period 1 and at the end of periods 1, 2, and 3. The effectiveness of different MMFS dosages on cognition, mood, and sleep quality will be assessed using a Neuropsychological Test Battery, Profile of Mood States-Brief Form, daily sleep diaries, and Insomnia Severity Index. The safety profile of different MMFS dosages will be determined by monitoring the AE/SAE and subjective remarks during the study period. A range of safety and tolerability assessments will also be performed (including vital signs and laboratory tests).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged 60 to 85 inclusive at the time of screening with informed consent.
2. Subjects with body weight within 50 to 125 kg and height within 152.4 to 198.12 cm, able to comply with study requirements; have received high school diploma, GED, or equivalent.
3. Subjects must have regular access to an internet-connected computer, iPad, tablet computer, and/or smart phone to complete online assessments.
4. Subjects with difficulty in maintaining sleep by the following criteria:

   * Insomnia Severity Index (ISI) score ≥ 10 and ≤ 21

     * 2 (moderate) or greater on question 2 OR question 3 of ISI
5. Subjects with at least "moderate" neuropsychiatric symptoms, as determined by a score of 6 or higher on the Mild Behavioral Impairment - Checklist (MBI-C) informant-report scale;

   * Subjective report of worsened neuropsychiatric symptoms (e.g., MBI-C items such as motivation, depression, anxiety, impulse control, delusions) since age 50, with recent decline
6. Score ≤ 7 and ≥ 4 on the D-KEFS Trail Making Test Condition 4 - letter-number switching test of executive function at screening, controlled for motor speed (condition 5)

   * Subjective report of worsened memory since age 50, with recent decline
7. Score of ≤ 7 and ≥ 4 on WMS-IV Logical Memory II (Delayed)
8. Subjects must be fluent in English
9. Subject must be willing to submit to blood draw(s).
10. Subjects must be able to understand the study, agree to the requirements and restrictions, be able to attend all scheduled visits, and be willing to give voluntary consent to participate in the study.

Exclusion Criteria:

1. Subject with insomnia due to bladder problems, or other confounding medical condition such as chronic pain syndromes, chronic migraine, cardiac disease, nocturia (> 3 times/night), asthma, gastroesophageal reflux disease (GERD), or hot flashes, determined by investigators.
2. Subject diagnosed with severe sleep apnea that is not treated/well-managed (e.g., by regular use of Continuous Positive Airway Pressure, CPAP, or Bilevel Positive Airway Pressure, BIPAP, device)
3. Subject's residence is an institutional facility such as a nursing home.
4. Females of child-bearing potential as defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
5. History or diagnosis of any of the following sleep conditions:

   * Narcolepsy
   * Cataplexy (familial or idiopathic)
   * Circadian Rhythm Sleep Disorder
   * Primary Hypersomnia
6. Subjects with history or presence of any clinically significant cardiovascular (myocardial infarction; coronary angioplasty or bypass graft(s); valvular disease or repair; unstable angina pectoris; transient ischemic attack (TIA); cerebrovascular accidents (CVA); congestive heart failure or coronary artery disease (CAD), clinically important carotid or vertebrobasilar stenosis or plaque, pulmonary, respiratory, hepatic, renal (including poor kidney function, eGFR <55 mL/min), hematological (sickle cell anemia or thalassemia, sideroblastic anemia or anemia of any etiology), gastrointestinal, endocrine (diabetes type I or II), immunologic, dermatologic, neurological, psychiatric disease or disorder within 6 months, or any uncontrolled medical illness which in the opinion of the Investigator would jeopardize the safety of the subject.

   Nonetheless, subjects with controlled co-morbid conditions (including diabetes, hypertension, heart disease, etc.) are permitted if considered stable within three months of the study start. All concomitant medications, supplements, or other substances must be at stable doses for at least 3 months prior to screening and must be kept as stable as medically possible during the trial.
7. Any of the following based on clinician interview :

   1. Clinically significant psychiatric illness in past 6 months requiring hospitalization
   2. Other psychiatric condition that, in the investigator's opinion, would interfere with the subject's ability to participate in the study
8. Suicidal ideation with intent, with or without a plan or method in the past 1 month or suicidal behavior in the past 6 months of Screening
9. History of alcoholism or drug dependency/abuse within the last 5 years of Screening, according to interview
10. Recent history (within the 6 months prior to Screening) of regular consumption (3 or more days per week) of either:

    1. 2 or more (women) or 3 or more (men) alcoholic beverages per day or alcohol consumption within 3 hours prior to bedtime
    2. More than 600 mg caffeine a day (e.g., 4 standard 8-ounce cups of brewed coffee, or typically consumes caffeine after 4pm [16:00])
11. Known hypersensitivity to magnesium or to any of the formulation components (not including the common laxative effects of magnesium supplements)
12. Currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent, or intent to participate in another clinical trial at any time during the conduct of this trial
13. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Test Battery (NTB; computerized, at home, on-line) composite score | 2 weeks each dose
  NTB consists of 5 cognitive tests, including: 1) N-Back Test for working memory; 2) Trail Making Test (TMT) assessing psychomotor processing speed and cognitive flexibility; 3) Backwards Digit Span Test for working memory; 4) Digit Symbol Substitution Test (DSST) measuring psychomotor processing speed; and 5) Block Tapping Test assessing visuo-spatial working memory. For each test, scores will be normalized using a z-score transformation. The mean of the 5 z-scores for each subject will be compared between low dose MMFS, high dose MMFs, and placebo groups. A score of 0 designates average performance. Each point above 0 designates 1 standard deviation above average and each point below 0 designates 1 standard deviation below average.

SECONDARY OUTCOMES:
Total Mood Disturbance (TMD) composite score measured by the Profile of Mood States - Brief Form (POMS-BF) | 2 weeks each dose, mean of days 3-7 of week 2 in each of the 3 periods
  POMS-BF is a self-rated questionnaire on different moods over the past day. It consists of 30 questions pertaining to 6 domains of mood. Each question is rated on a 5-point scale (0-4). Lower scores indicate a better mood state. Comparison of the mean score between low dose MMFS, high dose MMFs, and placebo groups.
Consensus Sleep Diary for Morning - Subjective Sleep Quality | 2 weeks each dose, mean of days 3-7 of week 2 in each of the 3 periods
  Subjective measurements of daily anxiety by recording a daily diary (recorded in the morning) on a 10 point scale (1-10) with 1=Extremely poor and 10=Extremely good. Adapted from Consensus Sleep Diary.
Consensus Sleep Diary for Morning - Refreshed Feeling | 2 weeks each dose, mean of days 3-7 of week 2 in each of the 3 periods
  Subjective measurements of daily anxiety by recording a daily diary (recorded in the morning) on a 10 point scale (1-10) with 1=Extremely unrefreshed and 10=Extremely refreshed. Adapted from Consensus Sleep Diary.
Consensus Sleep Diary for Evening - Subjective Anxiety | 2 weeks each dose, mean of days 3-7 of week 2 in each of the 3 periods
  Subjective measurements of daily anxiety by recording a daily diary (recorded in the evening) on a 10 point scale (1-10) with 1=Extremely anxious and 10=Extremely relaxed. Adapted from Consensus Sleep Diary.
Consensus Sleep Diary for Evening - Subjective Depression | 2 weeks each dose, mean of days 3-7 of week 2 in each of the 3 periods
  Subjective measurements of daily anxiety by recording a daily diary (recorded in the evening) on a 10 point scale (1-10) with 1=Extremely depressed and 10=Extremely cheerful. Adapted from Consensus Sleep Diary.
Consensus Sleep Diary for Evening- Subjective Cognitive Ability | 2 weeks each dose, mean of days 3-7 of week 2 in each of the 3 periods
  Subjective measurements of daily anxiety by recording a daily diary (recorded in the evening) on a 10 point scale (1-10) with 1=Extremely poor and 10=Extremely good. Adapted from Consensus Sleep Diary.

OTHER OUTCOMES:
Insomnia Severity Index (ISI) score | 2 weeks each dose
  A self-rated questionnaire to assess the severity of insomnia in subjects. It has a total of 7 questions; each rated on a 5-point scale (0-4) with 4 being the worst. All of the scores will be added and the total score of ISI will be the outcome measure. The scores will be compared between each MMFS formulation week (MMFS low dose vs high) and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Burkindine, MD, Principal Investigator — Bio-Kinetic Clinical Applications, LLC
Locations (1):
- Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No